CLINICAL TRIAL: NCT04421118
Title: Study on The Precise Selection of Stent Diameter for Portal Hypertension Patients With Transjugular Intrahepatic Portosystemic Shunt Based on Computational Fluid Dynamics
Brief Title: The Precise Selection of Stent Diameter for Portal Hypertension Patients With TIPS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: LanZhou University (Other)
Responsible Party: Sponsor
Other Study IDs: HEPIC2002
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Compensated Advanced Chronic Liver Disease; Portal Hypertension
Keywords: Transjugular intrahepatic portosystemic shunt; Stent selection; Fluid dynamics simulation
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- standard portal pressure gradient measurement and CT scan: Procedure/Surgery:
  Portal pressure gradient measurement and CT imaging examination. Three-dimensional models reconstructing and fluid dynamics simulation.
  Interventions: Other: a non-invasive technology to evaluate hepatic venous pressure gradient and portal pressure gradient

INTERVENTIONS:
Other: a non-invasive technology to evaluate hepatic venous pressure gradient and portal pressure gradient — a non-invasive technology to evaluate hepatic venous pressure gradient and portal pressure gradient based on three-dimensional modeling and fluid dynamics simulation

SUMMARY:
The precise planning of TIPS, especially individual selection of stent diameter, is a hot and difficult topic in the field. We have successfully developed a non-invasive technology to evaluate hepatic venous pressure gradient and portal pressure gradient based on three-dimensional modeling and fluid dynamics simulation. We propose the concept of virtual stent-based portal pressure gradient for the first time. With invasive pressure as reference, the accuracy of virtual stent-based portal pressure gradient will be evaluated in levels of animal experiments and clinical trials. The predictive value of virtual stent-based portal pressure gradient for individualized selection of TIPS stent diameter will be further assessed.

DETAILED DESCRIPTION:
Transjugular intrahepatic portosystemic shunt (TIPS) is an effective treatment for portal hypertension related variceal bleeding. The precise planning of TIPS, especially individual selection of stent diameter, is a hot and difficult topic in the field. A stent with smaller diameter cannot effectively reduce portal pressure, and a stent with larger diameter might cause hepatic encephalopathy resulted from excessive blood shunt. Therefore, individualized selection of TIPS stent diameter closely correlates with intervention effect and clinical outcomes. In our previous study, we have successfully developed a non-invasive technology to evaluate hepatic venous pressure gradient and portal pressure gradient based on three-dimensional modeling and fluid dynamics simulation. In this project, we propose the concept of virtual stent-based portal pressure gradient for the first time. Accurate three-dimensional models of hepatic-portal vein system with stents of different diameters will be reconstructed using imaging control and modeling software. In addition, a standard procedure of fluid dynamics simulation will be fixed with the platform of finite element calculation. With invasive pressure as reference, the accuracy of virtual stent-based portal pressure gradient will be evaluated in levels of animal experiments and clinical trials. Lastly, the predictive value of virtual stent-based portal pressure gradient for individualized selection of TIPS stent diameter will be further assessed.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* age 18-75 years;
* high-risk treatment failure (e.g.Child-Pugh C or B grade with variceal bleeding);
* conventional drugs and endoscopic treatment of esophageal variceal bleeding are not good;
* End-stage liver disease with variceal bleeding before liver transplantation;
* successful implementation of TIPS;
* good compliance with the requirements formulated by the study;
* with written informed consent.

Exclusion Criteria:

* Liver transplantation in the past or planning liver transplantation in the 6 months;
* Common TIPS contraindications (e.g.NYHA level 2 of congestive heart failure ,history of pulmonary hypertension, portal vein trunk thrombosis, multiple liver cysts,or intrahepatic bile duct dilatation);
* severe liver dysfunction: prothrombin activity <40% or bilirubin> 50μmol / L or Child-Pugh score> 12;
* history of hepatic encephalopathy;
* serum creatinine> 133μmol / L;
* severe hyponatremia (blood sodium <125mmol / L);
* uncontrollable infections;
* allergic to intravenous contrast agent;
* subject refused to participate in the trial or without the ability to participate in informed consent;
* previous history of TIPS treatment;
* any comorbidities or conditions that affect the test results as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with compensated advanced chronic liver disease
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Accuracy of vsPPG | 1 day
  To assess the accuracy of vsPPG at the clinical level(virtual PPG values and real PPG value)

SECONDARY OUTCOMES:
Guiding value of vsPPG | 1 day
  To assess the Guiding value of vsPPG at the level of animal experiments(the predictive value of virtual stent-based portal pressure gradient for individualized selection of TIPS stent diameter)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-hui Sun, MD,PH.D, Study Director — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Qi X, Li Z, Huang J, Zhu Y, Liu H, Zhou F, Liu C, Xiao C, Dong J, Zhao Y, Xu M, Xing S, Xu W, Yang C. Virtual portal pressure gradient from anatomic CT angiography. Gut. 2015 Jun;64(6):1004-5. doi: 10.1136/gutjnl-2014-308543. Epub 2014 Nov 14. No abstract available. PMID 25398771
- [Background] Qi X, An W, Liu F, Qi R, Wang L, Liu Y, Liu C, Xiang Y, Hui J, Liu Z, Qi X, Liu C, Peng B, Ding H, Yang Y, He X, Hou J, Tian J, Li Z. Virtual Hepatic Venous Pressure Gradient with CT Angiography (CHESS 1601): A Prospective Multicenter Study for the Noninvasive Diagnosis of Portal Hypertension. Radiology. 2019 Feb;290(2):370-377. doi: 10.1148/radiol.2018180425. Epub 2018 Nov 20. PMID 30457484
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Mokdad AA, Lopez AD, Shahraz S, Lozano R, Mokdad AH, Stanaway J, Murray CJ, Naghavi M. Liver cirrhosis mortality in 187 countries between 1980 and 2010: a systematic analysis. BMC Med. 2014 Sep 18;12:145. doi: 10.1186/s12916-014-0145-y. PMID 25242656
- [Background] Estes C, Anstee QM, Arias-Loste MT, Bantel H, Bellentani S, Caballeria J, Colombo M, Craxi A, Crespo J, Day CP, Eguchi Y, Geier A, Kondili LA, Kroy DC, Lazarus JV, Loomba R, Manns MP, Marchesini G, Nakajima A, Negro F, Petta S, Ratziu V, Romero-Gomez M, Sanyal A, Schattenberg JM, Tacke F, Tanaka J, Trautwein C, Wei L, Zeuzem S, Razavi H. Modeling NAFLD disease burden in China, France, Germany, Italy, Japan, Spain, United Kingdom, and United States for the period 2016-2030. J Hepatol. 2018 Oct;69(4):896-904. doi: 10.1016/j.jhep.2018.05.036. Epub 2018 Jun 8. PMID 29886156
- [Background] Trebicka J, Bastgen D, Byrtus J, Praktiknjo M, Terstiegen S, Meyer C, Thomas D, Fimmers R, Treitl M, Euringer W, Sauerbruch T, Rossle M. Smaller-Diameter Covered Transjugular Intrahepatic Portosystemic Shunt Stents Are Associated With Increased Survival. Clin Gastroenterol Hepatol. 2019 Dec;17(13):2793-2799.e1. doi: 10.1016/j.cgh.2019.03.042. Epub 2019 Mar 30. PMID 30940552